CLINICAL TRIAL: NCT02190032
Title: Comparison of Individually Modified Angled Tube and Conventional Angled Tube in Double-lumen Endotracheal Tube Intubation: A Randomized Clinical Trial
Brief Title: Modified Angled Tube vs. Conventional Angled Tube in Double-lumen Endotracheal Tube Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2014-06-003-004
Record Dates: First submitted 2014-07-06; First posted 2014-07-15 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Intubation, Intratracheal; Thoracic Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Intubating a manufacturer-provided-angled double-lumen tube (=Conventional-angled group,"MallinckrodtTM endotracheal tube", Covidien)
  Interventions: Device: Mallinckrodt endobronchial tube with a conventional angle
- Tube angle modification (Experimental): The angle of the double lumen tube(MallinckrodeTM endotracheal tube) is modified individually.At sniffing position, the distal tip of the tube is placed at the patient's cricoid cartilage level and the tube is bent at the intersection point of the two airway axes (oropharyngeal axis and tracheal axis) with an angle between the two axes.
  Interventions: Device: Mallinckrodt endotracheal tube with a modified angle

INTERVENTIONS:
Device: Mallinckrodt endotracheal tube with a modified angle — At sniffing position, the distal tip of a double-lumen tube is located at the patient's cricoid cartilage level and then the tube is bent at the intersection point of oral axis and the pharyngolaryngeal axis with an angle between the two axes.
  Other Names: Tube angle modification; ("MallinckrodeTM endotracheal tube", Covidien)
  Arms: Tube angle modification
Device: Mallinckrodt endobronchial tube with a conventional angle — Inserting a manufacturer-provided conventional-angled tube
  Other Names: Mallinckrodt endobronchial tube, Covidien, with conventional-angled tube
  Arms: Control group

SUMMARY:
The investigators are trying to compare the individually modified-angled tube and the conventional-angled tube in ease of double lumen endotracheal tube insertion and the incidence of related postoperative complications.

DETAILED DESCRIPTION:
Inserting a double lumen endotracheal tube is somewhat more difficult than a single lumen tube intubation because of its larger outer diameter and the more rigid feature. Moreover, the airway axes (oral-,pharyngeal-, and laryngotracheal axis) are not always straight under sniffing condition. Therefore, to make easy to insert a double-lumen tube and reduce the tube-related complications, we are trying to compare the individually angle-modified tube and the manufacturer-provided-angled tube.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing thoracic surgery under one lung ventilation
* Subjects older than 20 yrs who can give written informed consent

Exclusion Criteria:

* Those who need rapid sequence intubation
* Those with cervical spinal disease (cervical spinal injury, rheumatoid arthritis with atlantoaxial subluxation)
* Those with oropharyngeal obstructive disease (including tumor, foreign body)
* Those who are expected prolonged intubation after surgery
* Those who are pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The time taken to intubate a double-lumen tube | within 60 sec
  The time taken to insert the tube begins when the laryngoscope passes the patient's lips and ends when the tube passes the vocal cords

SECONDARY OUTCOMES:
The number of attempts needed for successful intubation | Intubation
The time taken for the first attempt of intubation | within 60 sec
Postoperative sore throat, hoarseness or dysphagia | 30 minutes and 24hours after extubation

OTHER OUTCOMES:
Hemodynamic change | 1, 3 and 5 min after intubation
  We will record patient's heart rate, blood pressure and any used cardiovascular drugs at 1, 3 and 5 min after intubation
Intubation difficulty scale score | At intubation
  Intubation difficulty Scale score is a function of seven parameters : number of attempts, number of operators, number of alternative techniques, cormack grade, lifting force needed, laryngeal pressure and vocal cord mobility.
  (Ref: Intubation Difficulty Scale, Anesthesiology 1997;87:1290-7)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hwan Lee, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Min JJ, Lee JH, Kang SH, Kim E, Lee SM, Cho JH, Kim HK. The Fast and Easy Way for Double-Lumen Tube Intubation: Individual Angle-Modification. PLoS One. 2016 Aug 18;11(8):e0161434. doi: 10.1371/journal.pone.0161434. eCollection 2016. PMID 27537372